CLINICAL TRIAL: NCT00935688
Title: An Examination of ACT Strategy in South-central Asia on Falciparum Malaria in a Context Where Vivax is the Major Species
Brief Title: Examination of ACT Implementation in a Vivax / Falciparum Co-endemic Area
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Health Protection and Research Organisation (Unknown); HealthNet TPO (Other); Medical Emergency Relief International (Merlin) (Unknown)
Responsible Party: Principal Investigator, Mark Rowland, Principle Investigator, Professor of Entomology and Malaria Control, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ACT Consortium
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Malaria; Fever
Keywords: malaria; rapid diagnostic tests; afghanistan; Non-specific fever
MeSH Terms: conditions — Malaria; Fever | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rapid diagnostic tests (Experimental): malaria diagnosis by rapid diagnostic test
  Interventions: Other: Rapid diagnostic test
- Clinic Microscopy (No Intervention): malaria diagnosed with field light-microscopy
- Clinical Diagnosis (No Intervention): Malaria diagnosed on the basis of clinical symptoms alone (i.e. not laboratory diagnosis)

INTERVENTIONS:
Other: Rapid diagnostic test — Dual species test for P. vivax and P. falciparum malaria
  Arms: Rapid diagnostic tests

SUMMARY:
In areas of which are co-endemic for vivax and falciparum malaria, treatments for the two diseases often differ and this may lead to mistreatment. This places an emphasis on diagnosis at the health service provision level. Diagnosis is also important when malaris endemicity is low - most fevers are not caused by disease. These two issues mean that most malaria and fevers are not adequately treated, even though the drugs may be effective; many patients who do not have malaria are treated for the disease, and patients with malaria may get the wrong treatment for their species. The study aims to test the effectiveness of employing rapid diagnostic tests and will study the effect on correct treatment.

DETAILED DESCRIPTION:
The study will randomly assign diagnostic methods, either with clinical diagnosis, field microscopy or rapid diagnostic tests. The study will take place in 22 clinics in Eastern and Northern Afghanistan, both areas with low transmission of predominantly vivax malaria. They differ in their locations and their current standard diagnostic methods.

The study will examine the result of the diagnostic test in the clinic against the result of reference slides and PCR to estimate the number of cases correctly treated in each arm. This will be a measure of the effectiveness of diagnosis (and the physicians response to the diagnosis) and be influential in considering modalities for diagnostic delivery

ELIGIBILITY:
Inclusion Criteria:

* Any patient where the clinician* considers malaria in the diagnosis - either prescribing an antimalarial or would request a malaria test if available or referring for diagnosis of malaria elsewhere.
* Patient, or parent/guardian, gives informed consent to the study.

Exclusion Criteria:

* Patients with a result from another facility
* Patients referred on for diagnosis in the private sector
* Patients the clinician decides to treat presumptively without requesting a test (defined as treating prior to randomisation)
* Where the clinician requests microscopy specifically due to clinical need prior to randomisation will not be randomised in the trial, but will be noted as part of the study and a reference slide and clinical information will be taken following consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4200 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients correctly treated | 2009-2010
  Composite measure defined as patients with Pf malaria receiving ACT Drugs; Pv malaria receiving CQ; patients with no malaria receiving no antimalarial drugs.
  NOTE: Previously reported here as "Proportion of patients incorrectly treated" being 1 minus the Proportion correctly treated. No change in how the outcome was measured.

SECONDARY OUTCOMES:
% of PV patients not receiving CQ % of PF patients not receiving SP/AS | 2009-2010
Diagnostic Accuracy of the different malaria tests | 2009-2010
  Sensitivity and specificity of mRDTs, Microscopy and clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Toby Leslie, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Afghanistan (2):
  - Merlin, Kunduz, Kunduz
  - HealthNet TPO, Jalalabad, Nangarhar

REFERENCES:
- [Derived] Hansen KS, Grieve E, Mikhail A, Mayan I, Mohammed N, Anwar M, Baktash SH, Drake TL, Whitty CJ, Rowland MW, Leslie TJ. Cost-effectiveness of malaria diagnosis using rapid diagnostic tests compared to microscopy or clinical symptoms alone in Afghanistan. Malar J. 2015 May 28;14:217. doi: 10.1186/s12936-015-0696-1. PMID 26016871
- [Derived] Leslie T, Mikhail A, Mayan I, Cundill B, Anwar M, Bakhtash SH, Mohammed N, Rahman H, Zekria R, Whitty CJ, Rowland M. Rapid diagnostic tests to improve treatment of malaria and other febrile illnesses: patient randomised effectiveness trial in primary care clinics in Afghanistan. BMJ. 2014 Jun 19;348:g3730. doi: 10.1136/bmj.g3730. PMID 24948695